CLINICAL TRIAL: NCT04669340
Title: E-learning in Patient Education to Patients With Rheumatoid Arthritis - An Evaluation of the Effectiveness, the Patient Perspective and the Implementation
Brief Title: E-learning in Patient Education to Patients With Rheumatoid Arthritis
Acronym: WEB-RA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: Randers Regional Hospital (Other); Aalborg University Hospital (Other); Horsens Hospital (Other); TrygFonden, Denmark (Industry); Novo Nordisk A/S (Industry); Regionshospital Nordjylland (Other Government)
Responsible Party: Principal Investigator, Line Raunsbæk Knudsen, Nurse, PhD student, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1-16-02-52-19
Record Dates: First submitted 2020-11-27; First posted 2020-12-16 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Rheumatoid Arthritis; Patient Involvement; Self Efficacy
Keywords: Patient education; Self-management; Technology; E-learning
MeSH Terms: conditions — Arthritis, Rheumatoid; Patient Participation

STUDY DESIGN:
Masking Description: Masking not possible due to mode of intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants in the intervention group will receive patient education through an e-learning program at home. A study nurse will introduce patients to the program and they will be asked to accomplish the program within four weeks. Furthermore, they will be encouraged to go through the program as many times as necessary and involve family and relatives if they like.
  Both groups will receive one planned phone call regarding medication 2-3 weeks after they started taking the medicine. Furthermore, both groups will be referred to a physiotherapist if needed. All patients have access to contact the out-patient clinic as needed throughout the study period.
  Interventions: Other: E-learning patient education
- Control group (Active Comparator): Participants in the control group will receive conventional patient education from a nurse in the out-patient clinic within four weeks after inclusion. Relatives can take part in the conversation.
  Both groups will receive one planned phone call regarding medication 2-3 weeks after they started taking the medicine. Furthermore, both groups will be referred to a physiotherapist if needed. All patients have access to contact the out-patient clinic as needed throughout the study period.
  Interventions: Other: Standard face-to-face patient education

INTERVENTIONS:
Other: E-learning patient education — The intervention implies patient education through an e-learning program. The program consists of three learning modules covering knowledge of rheumatoid arthritis, medication, examinations, complications and daily living with RA. Module 1 consists of 'need to know' information about disease management, symptoms and medication. Thus, it is mandatory and must be completed before entering module 2 and 3. In module 2 and 3, patients can move around on the basis of their individual needs.
  The duration of the full program is approximately two hours, but may vary dependent on the individual user needs. The program may be used as much as needed throughout the study period.
  Arms: Intervention group
Other: Standard face-to-face patient education — The intervention implies usual care, i.e. face-to-face patient education in a one-hour session with a nurse at the hospital. This form of patient education is based on the patients individual need for information and guidance in relation to rheumatoid arthritis and medication. Thus, aspects of daily life with the disease is discussed at the beginning and forms the conversation. However, as a standard, information of the disease, disease management, symptoms and medication must be discussed with the patient and relatives.
  Arms: Control group

SUMMARY:
Rheumatoid arthritis (RA) is a chronic inflammatory disease that primarily causes pain, swelling and stiffness in the joints. The disease may reduce normal functioning and thereby quality of life.

Patient education (PE), with the aim of supporting patients to self-manage their disease is an important part of the treatment and care to patients with RA. PE supports people in living with RA by offering knowledge of the disease, symptoms and treatment as well as guidance in coping with the disease in everyday life. In recent years, the number of people with RA has risen and in general people lives longer. This places new demands on the healthcare system for alternatives to conventional care, e.g. through web technology and remote care.

Often PE is provided through face-to-face interactions with health professionals at the hospital and thus far, only a small number of studies have been conducted within the area of web-based PE targeting people with RA. A few studies within RA and other chronic diseases shows that online tools and online educational programs may enhance patient's knowledge of the disease and treatment and improve self-management and quality of life.

Internet and technology is a great part of everyday life, however, variation is seen in computer skills and likewise in health literacy skills.

Even so, PE based on web technology may have several advantages, e.g. the accessibility and the possibility to seek for information as needed and repeatedly in familiar surroundings and possibly with relatives.

Moreover, the integration of words and images can promote deeper understanding and learning since both auditory and visual channels are used. Possible disadvantages may be related to the absence of face-to-face contact with healthcare professionals.

Given the need for alternative solutions to the conventional face-to-face contact, the investigators have developed an e-learning program targeting newly diagnosed patients with RA. The purpose of the program is to support self-management of the disease. The program takes into consideration peoples different competencies and assumptions by presenting information in an easy, inspiring and entertaining way. The program consists of three learning modules covering knowledge of the disease, medication, examinations, complications and daily living with RA, e.g. coping with emotions, pain, fatigue, physical activity, work etc.

In keeping with different ways of learning and to support people's different competencies, the program offers a combination of animations, graphics, videos, podcasts, quizzes, written text and spoken words.

Given the limited evidence about the effectiveness of web-based PE in RA, the intention behind the study is to evaluate the e-learning program.

The project will be divided into three parts. In the first part the effect of the e-learning program will be evaluated. Approximately 200-230 patients from four rheumatology clinics in Denmark will be included. Half of the participants will receive education at home through the e-learning program and the other half will receive conventional education at the hospital.

The effect of PE will be evaluated through questionnaires covering self-efficacy, knowledge of RA and medication, medication taking, health literacy skills and quality of life. Additionally, disease activity, physical functioning, pain and fatigue will be measured.

Furthermore, the investigators will examine the use of the e-learning program, such as time consumption and completed modules. Finally, telephone contacts from patients to the outpatient clinics will be measured to investigate possible causal relationships between the information provided through PE and the need for additional information or guidance related to self-management. The number of out-patient visits in the clinic will also be measured.

In the second part the investigators will explore the perceptions of receiving PE through the e-learning program from the perspective of patients with RA. This will be explored through individually interviews with approximately 20-25 patients.

In the third part the complexities in the e-learning program to improve chances of success in implementation of the technology in clinical practice, i.e. outside the project, will be explored. Through focus group interviews with nurses and doctors involved in the project, the investigators will explore perspectives of using the program. The interviews will be based on a framework covering both successes, challenges and failures in relation to the technology, the patient group, values and the organisation.

Furthermore, the investigators will revisit the patient interviews from the second part in order to obtain information about these aspects from the patient perspective.

The investigators hypothesize that the e-learning PE program will be superior to standard face-to-face PE in improving self-efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid arthritis according to the American College of Rheumatology 2010 criteria within the past 3 - 4 months (before inclusion)
* Able to speak and understand Danish
* Able to access the Internet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Change in self-efficacy from baseline after 1, 3, 6 and 12 months | 1, 3, 6 and 12 months
  The primary outcome is the Danish version of the rheumatoid arthritis self-efficacy questionnaire (RASE). This is used as the primary outcome as self-efficacy is considered a pre-condition of self-management and as RASE is developed specifically for measuring self-efficacy in rheumatoid arthritis.

SECONDARY OUTCOMES:
Change in knowledge of RA from baseline after 1, 3, 6 and 12 months | 1, 3, 6 and 12 months
  Knowledge of RA will be measured through the PKQ-RA (Patient knowledge questionnaire - Rheumatoid arthritis) questionnaire. Ahead of this study we have translated, validated and adapted this questionnaire into a Danish Version reflecting the content of our e-learning program and updated this to reflect current treatment guidelines.
Change in compliance from baseline after 1, 3, 6 and 12 months | 1, 3, 6 and 12 months
  The 5 item compliance questionnaire (CQR5) will be used to measure patients adherence to medication.
Change in health literacy from baseline after 1, 3, 6 and 12 month | 1, 3, 6 and 12 months
  Parts of the health literacy questionnaire (HLQ) will be used. A set of abilities, such as reading and acting upon written health information, communicating needs to health professionals, and understanding health instructions is measured through this instrument.
Change in health-related quality of life from baseline after 1, 3, 6 and 12 months | 1, 3, 6 and 12 months
  Quality of life will be measured through the EQ-5D (European Quality of Life - 5 Dimensions) questionnaire which covers mobility, personal care, usual activities, pain, anxiety and depression.

CONTACTS AND LOCATIONS:
Overall Officials: Line R Knudsen, RN, MCN, Principal Investigator — Aarhus University Hospital and Aarhus University
Locations (5):
- Denmark (5):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus N
  - Hjørring Regional Hospital, Hjørring
  - Horsens Hospital, Horsens
  - Randers Regional Hospital, Randers

IPD SHARING:
Plan to Share IPD: Yes
We intend to publish the study protocol in an international peer reviewed journal.
Supporting Information: Study Protocol
Time Frame: At the beginning of 2021.

REFERENCES:
- [Background] Brady TJ, Murphy L, O'Colmain BJ, Beauchesne D, Daniels B, Greenberg M, House M, Chervin D. A meta-analysis of health status, health behaviors, and health care utilization outcomes of the Chronic Disease Self-Management Program. Prev Chronic Dis. 2013;10:120112. doi: 10.5888/pcd10.120112. PMID 23327828
- [Background] Zangi HA, Ndosi M, Adams J, Andersen L, Bode C, Bostrom C, van Eijk-Hustings Y, Gossec L, Korandova J, Mendes G, Niedermann K, Primdahl J, Stoffer M, Voshaar M, van Tubergen A; European League Against Rheumatism (EULAR). EULAR recommendations for patient education for people with inflammatory arthritis. Ann Rheum Dis. 2015 Jun;74(6):954-62. doi: 10.1136/annrheumdis-2014-206807. Epub 2015 Mar 3. PMID 25735643
- [Background] Cross M, Smith E, Hoy D, Carmona L, Wolfe F, Vos T, Williams B, Gabriel S, Lassere M, Johns N, Buchbinder R, Woolf A, March L. The global burden of rheumatoid arthritis: estimates from the global burden of disease 2010 study. Ann Rheum Dis. 2014 Jul;73(7):1316-22. doi: 10.1136/annrheumdis-2013-204627. Epub 2014 Feb 18. PMID 24550173
- [Background] Minichiello E, Semerano L, Boissier MC. Time trends in the incidence, prevalence, and severity of rheumatoid arthritis: A systematic literature review. Joint Bone Spine. 2016 Dec;83(6):625-630. doi: 10.1016/j.jbspin.2016.07.007. Epub 2016 Sep 5. PMID 27616690
- [Background] Bech B, Primdahl J, van Tubergen A, Voshaar M, Zangi HA, Barbosa L, Bostrom C, Boteva B, Carubbi F, Fayet F, Ferreira RJO, Hoeper K, Kocher A, Kukkurainen ML, Lion V, Minnock P, Moretti A, Ndosi M, Pavic Nikolic M, Schirmer M, Smucrova H, de la Torre-Aboki J, Waite-Jones J, van Eijk-Hustings Y. 2018 update of the EULAR recommendations for the role of the nurse in the management of chronic inflammatory arthritis. Ann Rheum Dis. 2020 Jan;79(1):61-68. doi: 10.1136/annrheumdis-2019-215458. Epub 2019 Jul 12. PMID 31300458
- [Background] Lorig KR, Holman H. Self-management education: history, definition, outcomes, and mechanisms. Ann Behav Med. 2003 Aug;26(1):1-7. doi: 10.1207/S15324796ABM2601_01. PMID 12867348
- [Background] Lorig KR, Ritter P, Stewart AL, Sobel DS, Brown BW Jr, Bandura A, Gonzalez VM, Laurent DD, Holman HR. Chronic disease self-management program: 2-year health status and health care utilization outcomes. Med Care. 2001 Nov;39(11):1217-23. doi: 10.1097/00005650-200111000-00008. PMID 11606875
- [Background] Lorig KR, Sobel DS, Stewart AL, Brown BW Jr, Bandura A, Ritter P, Gonzalez VM, Laurent DD, Holman HR. Evidence suggesting that a chronic disease self-management program can improve health status while reducing hospitalization: a randomized trial. Med Care. 1999 Jan;37(1):5-14. doi: 10.1097/00005650-199901000-00003. PMID 10413387
- [Background] Holman H LK. Perceived self-efficacy in self-management of chronic disease. In: Schwarzer R, editor. Self-efficacy: Thought Control of Action. 1st ed. London: Taylor & Francis; 1994: 305-21
- [Background] Bandura A. Exercise of personal agency through the self-efficacy mechanism. In: Schwarzer R, editor. Self-efficacy: thought control of action. London: Taylor & Francis; 1994 (1st Ed.): 3-38.
- [Background] Conner M, Norman P. Predicting health behavior: Research and practice with social cognition models. Open University Press. New York. 2005
- [Background] Leventhal H, Brissette I, Leventhal EA. The common-sense model of self-regulation of health and illness. In: Cameron L.D., Leventhal H (Ed.). The self-regulation of health and illness behavior. Routledge. London. 2003.
- [Background] Leventhal H, Phillips LA, Burns E. The Common-Sense Model of Self-Regulation (CSM): a dynamic framework for understanding illness self-management. J Behav Med. 2016 Dec;39(6):935-946. doi: 10.1007/s10865-016-9782-2. Epub 2016 Aug 11. PMID 27515801
- [Background] Shigaki CL, Smarr KL, Siva C, Ge B, Musser D, Johnson R. RAHelp: an online intervention for individuals with rheumatoid arthritis. Arthritis Care Res (Hoboken). 2013 Oct;65(10):1573-81. doi: 10.1002/acr.22042. PMID 23666599
- [Background] Lorig KR, Ritter PL, Laurent DD, Plant K. The internet-based arthritis self-management program: a one-year randomized trial for patients with arthritis or fibromyalgia. Arthritis Rheum. 2008 Jul 15;59(7):1009-17. doi: 10.1002/art.23817. PMID 18576310
- [Background] Weymann N, Dirmaier J, von Wolff A, Kriston L, Harter M. Effectiveness of a Web-based tailored interactive health communication application for patients with type 2 diabetes or chronic low back pain: randomized controlled trial. J Med Internet Res. 2015 Mar 3;17(3):e53. doi: 10.2196/jmir.3904. PMID 25736340
- [Background] Lorig K, Ritter PL, Laurent DD, Plant K, Green M, Jernigan VB, Case S. Online diabetes self-management program: a randomized study. Diabetes Care. 2010 Jun;33(6):1275-81. doi: 10.2337/dc09-2153. Epub 2010 Mar 18. PMID 20299481
- [Background] Armstrong AW, Kim RH, Idriss NZ, Larsen LN, Lio PA. Online video improves clinical outcomes in adults with atopic dermatitis: a randomized controlled trial. J Am Acad Dermatol. 2011 Mar;64(3):502-7. doi: 10.1016/j.jaad.2010.01.051. Epub 2011 Jan 13. PMID 21236514
- [Background] Higgins O, Sixsmith J, Barry MM, Domegan C. A literature review on health information seeking behaviour on the web: a health consumer and health professional perspective. Stockholm: ECDC; 2011
- [Background] Sorensen K, Van den Broucke S, Fullam J, Doyle G, Pelikan J, Slonska Z, Brand H; (HLS-EU) Consortium Health Literacy Project European. Health literacy and public health: a systematic review and integration of definitions and models. BMC Public Health. 2012 Jan 25;12:80. doi: 10.1186/1471-2458-12-80. PMID 22276600
- [Background] Nariman HN. Soap Operas for Social Change - Toward a methodology for entertainment-education television. Praeger Publishers; 1993
- [Background] Mayer R. The Cambridge handbook of multimedia learning. 2005. New York
- [Background] Singhal A, Cody MJ, Rogers EM, Sabido M (editors). Entertainment-education and social change - History, research and practice. Taylor and Francis; 2003
- [Background] Lopez-Olivo MA, Ingleshwar A, Volk RJ, Jibaja-Weiss M, Barbo A, Saag K, Leong A, Suarez-Almazor ME. Development and Pilot Testing of Multimedia Patient Education Tools for Patients With Knee Osteoarthritis, Osteoporosis, and Rheumatoid Arthritis. Arthritis Care Res (Hoboken). 2018 Feb;70(2):213-220. doi: 10.1002/acr.23271. Epub 2017 Dec 29. PMID 28464546
- [Background] Funnel SC, Rogers PJ. Purposeful program theory. Effective use of theories of change and logic models. Jossey-Bass. San Francisco. 2011
- [Background] Morgan DL. Focus groups as qualitative research. 1997. Sage Publications, Inc. California
- [Background] Kristiansen TM, Primdahl J, Antoft R, Horslev-Petersen K. Everyday life with rheumatoid arthritis and implications for patient education and clinical practice: a focus group study. Musculoskeletal Care. 2012 Mar;10(1):29-38. doi: 10.1002/msc.224. Epub 2011 Dec 26. PMID 22213280
- [Background] Zuidema RM, Repping-Wuts H, Evers AW, Van Gaal BG, Van Achterberg T. What do we know about rheumatoid arthritis patients' support needs for self-management? A scoping review. Int J Nurs Stud. 2015 Oct;52(10):1617-24. doi: 10.1016/j.ijnurstu.2015.05.008. Epub 2015 Jun 9. PMID 26117711
- [Background] Radford S, Carr M, Hehir M, Davis B, Robertson L, Cockshott Z, Tipler S, Hewlett S. 'It's quite hard to grasp the enormity of it': perceived needs of people upon diagnosis of rheumatoid arthritis. Musculoskeletal Care. 2008 Sep;6(3):155-67. doi: 10.1002/msc.132. PMID 18649347
- [Background] Meesters JJ, Vliet Vlieland TP, Hill J, Ndosi ME. Measuring educational needs among patients with rheumatoid arthritis using the Dutch version of the Educational Needs Assessment Tool (DENAT). Clin Rheumatol. 2009 Sep;28(9):1073-7. doi: 10.1007/s10067-009-1190-3. Epub 2009 May 16. PMID 19449083
- [Background] Braun V, Clarke V. Using thematic analysis in psychology. Qualitative research in psychology. 2006; 3 (2): 77-101
- [Background] Elwyn G, Kreuwel I, Durand MA, Sivell S, Joseph-Williams N, Evans R, Edwards A. How to develop web-based decision support interventions for patients: a process map. Patient Educ Couns. 2011 Feb;82(2):260-5. doi: 10.1016/j.pec.2010.04.034. Epub 2010 Jun 2. PMID 20627644
- [Background] Fayers PM, Machin D. Quality of Life - The assessment, analysis and interpretation of patient-reported outcomes. 2007. John Wiley & Sons Ltd. England
- [Background] Collins D. Pretesting survey instruments: an overview of cognitive methods. Qual Life Res. 2003 May;12(3):229-38. doi: 10.1023/a:1023254226592. PMID 12769135
- [Background] Aletaha D, Neogi T, Silman AJ, Funovits J, Felson DT, Bingham CO 3rd, Birnbaum NS, Burmester GR, Bykerk VP, Cohen MD, Combe B, Costenbader KH, Dougados M, Emery P, Ferraccioli G, Hazes JM, Hobbs K, Huizinga TW, Kavanaugh A, Kay J, Kvien TK, Laing T, Mease P, Menard HA, Moreland LW, Naden RL, Pincus T, Smolen JS, Stanislawska-Biernat E, Symmons D, Tak PP, Upchurch KS, Vencovsky J, Wolfe F, Hawker G. 2010 Rheumatoid arthritis classification criteria: an American College of Rheumatology/European League Against Rheumatism collaborative initiative. Arthritis Rheum. 2010 Sep;62(9):2569-81. doi: 10.1002/art.27584. PMID 20872595
- [Background] Smolen JS, Landewe R, Bijlsma J, Burmester G, Chatzidionysiou K, Dougados M, Nam J, Ramiro S, Voshaar M, van Vollenhoven R, Aletaha D, Aringer M, Boers M, Buckley CD, Buttgereit F, Bykerk V, Cardiel M, Combe B, Cutolo M, van Eijk-Hustings Y, Emery P, Finckh A, Gabay C, Gomez-Reino J, Gossec L, Gottenberg JE, Hazes JMW, Huizinga T, Jani M, Karateev D, Kouloumas M, Kvien T, Li Z, Mariette X, McInnes I, Mysler E, Nash P, Pavelka K, Poor G, Richez C, van Riel P, Rubbert-Roth A, Saag K, da Silva J, Stamm T, Takeuchi T, Westhovens R, de Wit M, van der Heijde D. EULAR recommendations for the management of rheumatoid arthritis with synthetic and biological disease-modifying antirheumatic drugs: 2016 update. Ann Rheum Dis. 2017 Jun;76(6):960-977. doi: 10.1136/annrheumdis-2016-210715. Epub 2017 Mar 6. PMID 28264816
- [Background] Primdahl J, Wagner L, Horslev-Petersen K. Self-efficacy in rheumatoid arthritis: translation and test of validity, reliability and sensitivity of the Danish version of the Rheumatoid Arthritis Self-Efficacy Questionnaire (RASE). Musculoskeletal Care. 2010 Sep;8(3):123-35. doi: 10.1002/msc.172. PMID 20229609
- [Background] Primdahl J, Wagner L, Holst R, Horslev-Petersen K; AMBRA Study Group. The impact on self-efficacy of different types of follow-up care and disease status in patients with rheumatoid arthritis--a randomized trial. Patient Educ Couns. 2012 Jul;88(1):121-8. doi: 10.1016/j.pec.2012.01.012. Epub 2012 Mar 3. PMID 22386009
- [Background] Osborne RH, Batterham RW, Elsworth GR, Hawkins M, Buchbinder R. The grounded psychometric development and initial validation of the Health Literacy Questionnaire (HLQ). BMC Public Health. 2013 Jul 16;13:658. doi: 10.1186/1471-2458-13-658. PMID 23855504
- [Background] Maindal HT, Kayser L, Norgaard O, Bo A, Elsworth GR, Osborne RH. Cultural adaptation and validation of the Health Literacy Questionnaire (HLQ): robust nine-dimension Danish language confirmatory factor model. Springerplus. 2016 Aug 2;5(1):1232. doi: 10.1186/s40064-016-2887-9. eCollection 2016. PMID 27536516
- [Background] Hughes LD, Done J, Young A. A 5 item version of the Compliance Questionnaire for Rheumatology (CQR5) successfully identifies low adherence to DMARDs. BMC Musculoskelet Disord. 2013 Oct 8;14:286. doi: 10.1186/1471-2474-14-286. PMID 24103582
- [Background] Hurst NP, Kind P, Ruta D, Hunter M, Stubbings A. Measuring health-related quality of life in rheumatoid arthritis: validity, responsiveness and reliability of EuroQol (EQ-5D). Br J Rheumatol. 1997 May;36(5):551-9. doi: 10.1093/rheumatology/36.5.551. PMID 9189057
- [Background] Hennell SL, Brownsell C, Dawson JK. Development, validation and use of a patient knowledge questionnaire (PKQ) for patients with early rheumatoid arthritis. Rheumatology (Oxford). 2004 Apr;43(4):467-71. doi: 10.1093/rheumatology/keh069. Epub 2004 Jan 6. PMID 15024135
- [Background] Prevoo ML, van 't Hof MA, Kuper HH, van Leeuwen MA, van de Putte LB, van Riel PL. Modified disease activity scores that include twenty-eight-joint counts. Development and validation in a prospective longitudinal study of patients with rheumatoid arthritis. Arthritis Rheum. 1995 Jan;38(1):44-8. doi: 10.1002/art.1780380107. PMID 7818570
- [Background] Bruce B, Fries JF. The Stanford Health Assessment Questionnaire: a review of its history, issues, progress, and documentation. J Rheumatol. 2003 Jan;30(1):167-78. PMID 12508408
- [Background] Thorne S. Interpretive description: Qualitative Research for Applied Practice. New York and London: Routledge; 2016 (2ed).
- [Background] Greenhalgh T, Abimbola S. The NASSS Framework - A Synthesis of Multiple Theories of Technology Implementation. Stud Health Technol Inform. 2019 Jul 30;263:193-204. doi: 10.3233/SHTI190123. PMID 31411163
- [Background] Greenhalgh T, Wherton J, Papoutsi C, Lynch J, Hughes G, A'Court C, Hinder S, Fahy N, Procter R, Shaw S. Beyond Adoption: A New Framework for Theorizing and Evaluating Nonadoption, Abandonment, and Challenges to the Scale-Up, Spread, and Sustainability of Health and Care Technologies. J Med Internet Res. 2017 Nov 1;19(11):e367. doi: 10.2196/jmir.8775. PMID 29092808
- [Background] Greenhalgh T. How to improve success of technology projects in health and social care. Public Health Res Pract. 2018 Sep 27;28(3):2831815. doi: 10.17061/phrp2831815. PMID 30406256
- [Background] Abimbola S, Patel B, Peiris D, Patel A, Harris M, Usherwood T, Greenhalgh T. The NASSS framework for ex post theorisation of technology-supported change in healthcare: worked example of the TORPEDO programme. BMC Med. 2019 Dec 30;17(1):233. doi: 10.1186/s12916-019-1463-x. PMID 31888718
- [Derived] Knudsen LR, Ndosi M, Hauge EM, Lomborg K, Dreyer L, Aaboe S, Kjaer MB, Sorensen L, Volsmann L, Christensen HM, de Thurah A. Effectiveness of a novel digital patient education programme to support self-management of early rheumatoid arthritis: a randomized controlled trial. Rheumatology (Oxford). 2024 Sep 1;63(9):2547-2556. doi: 10.1093/rheumatology/keae177. PMID 38498833
- [Derived] Raunsbaek Knudsen L, Lomborg K, Ndosi M, Hauge EM, de Thurah A. The effectiveness of e-learning in patient education delivered to patients with rheumatoid arthritis: The WebRA study-protocol for a pragmatic randomised controlled trial. BMC Rheumatol. 2021 Dec 20;5(1):57. doi: 10.1186/s41927-021-00226-y. PMID 34924034
- See also: Statistics - The use of Internet in the Danish population — http://www.dst.dk/Site/Dst/Udgivelser/GetPubFile.aspx?id=20738&sid=itbef2016
- See also: Ten Attributes of Health Literate Health Care Organizations. Institute of Medicine - Of the national academies — http://nam.edu/wp-content/uploads/2015/06/BPH_Ten_HLit_Attributes.pdf

DOCUMENTS (1):
  • Study Protocol (2020-11-01): https://cdn.clinicaltrials.gov/large-docs/40/NCT04669340/Prot_000.pdf